CLINICAL TRIAL: NCT00288964
Title: Compassionate Use of the Hattler Respiratory Assist Catheter in Severe Respiratory Failure - A Clinical Trial
Brief Title: Use of the Hattler Respiratory Assist Catheter in Severe Respiratory Failure
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor no longer pursuing regulatory approval of investigational device
Sponsor: Alung Technologies (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 04/Q0104/125
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Emphysema; Acute Respiratory Distress Syndrome; Chronic Obstructive Pulmonary Disease; Asthma; Respiratory Insufficiency
Keywords: balloon; fiber; respiratory; oxygenator; Heart Failure; ARDS; COPD
MeSH Terms: conditions — Emphysema; Respiratory Distress Syndrome; Pulmonary Disease, Chronic Obstructive; Asthma; Respiratory Insufficiency; Heart Failure

INTERVENTIONS:
Device: Hattler Respiratory Assist Catheter

SUMMARY:
A new artificial lung device has been developed that potentially provides added support to mechanical ventilation for severely damaged lungs. The Hattler Respiratory Assist Catheter is designed to provide gas exchange (deliver oxygen and remove carbon dioxide) for a period of up to 7 days, providing more time for the lungs to improve.

Extrapolating from large animal data, the hypothesis is that the Hattler Catheter will be capable of providing 30% to 40% of the basal requirements of carbon dioxide exchange in a manner that is dependable and reproducible.

DETAILED DESCRIPTION:
The Hattler Catheter Respiratory Assist Device consists of a Catheter and a drive console. The catheter consists of a bundle of polypropylene hollow fibers (approximately 1000) in 30cm or 35cm length surrounding a helium filled balloon. The balloon is similar to an Intra-Aortic Balloon, however, it is pulsed at 300 beats per minute, while IABP typically operate at 120 bpm. The hollow fibers are similar to fibers utilized in external oxygenators for cardio-pulmonary bypass. No device exists on the market in which fibers surround a balloon, and no device exists on the market in which the hollow fiber bundle is designed to be inserted into the venous system, i.e., the vena cava. External oxygenators are designed to be used in an extracorporeal circulatory loop.

The Hattler Catheter drive console provides the power to drive the helium filled balloon while removing excess oxygen and carbon dioxide from the venous system via the catheter.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes, 18 years and older
* Have a terminally ill disease process
* On maximum ventilator support
* Intubated and unconscious
* Swan Ganz in place
* Hypoxic
* Unsuitable for organ donation

Exclusion Criteria:

* Circulatory shock (< 80 mmHg) and unresponsive to drug therapy and volume replacement
* Pregnancy
* Morbid obesity > 182 kg
* Weight < 41 kg
* History of bleeding disorders with contraindication to heparin
* Have a disease process with a contraindication to heparin
* Known internal jugular or femoral vein complications or abnormalities
* Known inferior vena cava (IVC) filter in place

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-11

PRIMARY OUTCOMES:
Effective insertion and removal as measured by hemostasis
Amount of effort required for both insertion and removal

SECONDARY OUTCOMES:
Peak gas exchange status within a maximum 7 day study

CONTACTS AND LOCATIONS:
Overall Officials: Steven Tsui, MD, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Trust, Papworth Everard, Cambridge, United Kingdom